CLINICAL TRIAL: NCT01376778
Title: A Randomized Trial to Prevent Congenital Cytomegalovirus (CMV)
Acronym: CMV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HD36801-CMV; U10HD036801 (NIH); U10HD027869 (NIH); U10HD027915 (NIH); U10HD034116 (NIH); U10HD034208 (NIH); U10HD040500 (NIH); U10HD040485 (NIH); U10HD040544 (NIH); U10HD040545 (NIH); U10HD040560 (NIH); U10HD040512 (NIH); U10HD053097 (NIH); U10HD068282 (NIH); U10HD068258 (NIH); U10HD068268 (NIH); UG1HD087230 (NIH); UG1HD087192 (NIH)
Record Dates: First submitted 2011-06-15; First posted 2011-06-20 (Estimated); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Congenital Cytomegalovirus Infection; Maternal Cytomegalovirus Infection
Keywords: Perinatology; Cytomegalovirus immune globulin; Cytogam; CMVIG infusions
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CMV hyperimmune globulin - Cytogam® (Active Comparator): Infusion of Cytogam®, Cytomegalovirus Immune Globulin Intravenous (Human) (CMV-IGIV)
  Interventions: Drug: CMV hyperimmune globulin
- Placebo (Placebo Comparator): IV 5% albumin diluted 1 to 9 with 5% Dextrose in water (D5W)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CMV hyperimmune globulin — The study's active drug is Cytogam® which is an immunoglobulin G (IgG) containing a standardized amount of antibody to CMV. This drug contains pooled adult human plasma selected for high titers of antibody for CMV, and is administered intravenously at a dose of 100 mg/kg body weight.
  Other Names: CMV-IGIV; Cytogam
  Arms: CMV hyperimmune globulin - Cytogam®
Other: Placebo — The matching placebo consists of AlbuRx® 5% diluted 1:9 with D5W. AlbuRx® 5% contains pooled adult human plasma.
  Arms: Placebo

SUMMARY:
Cytomegalovirus (CMV) is a common virus that usually presents with few if any side effects. When first infected, some people may have symptoms similar to mononucleosis (i.e., fatigue, weakness, fever, swollen glands). Most people in the United States are infected during childhood or as adults if they work around children. Pregnant women, who have not been infected with CMV in the past and become infected during pregnancy (i.e. a primary infection), may cause their babies to get infected with CMV. Babies that are infected may develop permanent disabilities including hearing loss and a small portion will die from the infection.

Currently it is not routine practice to screen pregnant women for CMV infection. Additionally, there is no agreement about how to evaluate and manage pregnant women infected with CMV for the first time. There is also no evidence that treatment is beneficial for the baby.

The purpose of this research study is to determine whether treating pregnant women who have a primary CMV infection with CMV antibodies will reduce the number of babies infected with CMV.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is the most common congenital infection, with approximately 44,000 congenitally infected infants in the U.S. per year. A substantial proportion of these infants will die or suffer permanent injury as a result of their infection. The severity of congenital infection is greatest with primary maternal CMV infection. Currently, there is no proven method of preventing congenital CMV infection, and the approach to primary maternal CMV infection in the United States is haphazard and ineffective. One small, non-randomized study suggests that maternal administration of CMV hyperimmune globulin may significantly reduce the rate of congenital CMV infection following maternal primary infection. The MFMU CMV Trial will address the primary research question: does maternal administration of CMV hyperimmune globulin lower the rate of congenital CMV infection among the offspring of women who have been diagnosed with primary CMV infection during early pregnancy?

The research study is funded by the Eunice Kennedy Shriver National Institutes of Child Health and Human Development (NICHD). Sixteen medical centers across the country are participating in this research study. In all, 800 pregnant women who are identified with a primary CMV infection will be enrolled in this research study. The children of these women will be evaluated and tested at one and two years of age.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary maternal CMV infection on the basis of one of the following:

  1. A positive CMV Immunoglobulin M (IgM) antibody and low-avidity maternal CMV Immunoglobulin G (IgG) antibody screen
  2. Evidence of maternal seroconversion with development of CMV IgG antibody following a prior negative CMV screen
* Gestational age at randomization no later than 23 weeks 6 days based on clinical information and evaluation of the earliest ultrasound; or no later than 27 weeks 6 days for women with a positive IgM, negative IgG initially screened before 23 weeks who are rescreened after 2-4 weeks and have evidence of IgG seroconversion.
* Singleton pregnancy. A twin pregnancy reduced to singleton (either spontaneously or therapeutically) before 14 weeks by project gestational age is acceptable.

Exclusion Criteria:

* Maternal CMV infection pre-dating pregnancy as defined by a high IgG avidity index or a positive IgG in the presence of a negative IgM.
* Known hypersensitivity to plasma or plasma derived products
* Planned termination of pregnancy
* Known major fetal anomalies or demise
* Maternal Immunoglobulin A (IgA) deficiency
* Planned use of immune globulin, ganciclovir, or valganciclovir
* Maternal renal disease (most recent pre-randomization serum creatinine ≥ 1.4 mg/dL; all women must have serum creatinine measured during the pregnancy and prior to randomization)
* Maternal immune impairment (e.g., HIV infection, organ transplant on anti-rejection medications)
* Findings on pre-randomization ultrasound suggestive of established fetal CMV infection (cerebral ventriculomegaly, microcephaly, cerebral or intra-abdominal calcifications, abnormalities of amniotic fluid volume, echogenic bowel or ascites). Abnormally low amniotic fluid volume is defined as no fluid prior to 14 weeks or maximum vertical pocket < 2 cm on or after 14 weeks gestation. Abnormally high amniotic fluid volume is defined as > 10 cm.
* Positive fetal CMV findings from culture (amniotic fluid) or PCR.
* Congenital infection with rubella, syphilis, varicella, parvovirus or toxoplasmosis diagnosed by serology and ultrasound or amniotic fluid testing.
* Intention of the patient or of the managing obstetricians for the delivery to be outside a Maternal-Fetal Medicine Units Network (MFMU) Network center
* Participation in another interventional study that influences fetal or neonatal death
* Unwilling or unable to commit to 2 year follow-up of the infant

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2012-04; Primary Completion 2019-10 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Longo, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Rebecca Clifton, PhD, Principal Investigator — George Washington University; Brenna Hughes, MD, Study Chair — Brown University
Locations (16):
- United States (16):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve-Metrohealth, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Magee Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas - Southwestern Medical Center, Dallas, Texas
  - University of Texas - Galveston, Galveston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The dataset will be shared per NIH policy after the completion and publication of the main analyses. Requests for datasets can be sent to mfmudatasets@bsc.gwu.edu.

REFERENCES:
- [Result] Hughes BL, Clifton RG, Rouse DJ, Saade GR, Dinsmoor MJ, Reddy UM, Pass R, Allard D, Mallett G, Fette LM, Gyamfi-Bannerman C, Varner MW, Goodnight WH, Tita ATN, Costantine MM, Swamy GK, Gibbs RS, Chien EK, Chauhan SP, El-Sayed YY, Casey BM, Parry S, Simhan HN, Napolitano PG, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A Trial of Hyperimmune Globulin to Prevent Congenital Cytomegalovirus Infection. N Engl J Med. 2021 Jul 29;385(5):436-444. doi: 10.1056/NEJMoa1913569. PMID 34320288
- [Result] Rouse DJ, Fette LM, Hughes BL, Saade GR, Dinsmoor MJ, Reddy UM, Pass R, Allard D, Mallett G, Clifton RG, Saccoccio FM, Permar SR, Gyamfi-Bannerman C, Varner MW, Goodnight WH, Tita ATN, Costantine MM, Swamy GK, Heyborne KD, Chien EK, Chauhan SP, El-Sayed YY, Casey BM, Parry S, Simhan HN, Napolitano PG, Macones GA; for the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network. Noninvasive Prediction of Congenital Cytomegalovirus Infection After Maternal Primary Infection. Obstet Gynecol. 2022 Mar 1;139(3):400-406. doi: 10.1097/AOG.0000000000004691. PMID 35115450
- [Derived] Dinsmoor MJ, Fette LM, Hughes BL, Rouse DJ, Saade GR, Reddy UM, Allard D, Mallett G, Thom EA, Gyamfi-Bannerman C, Varner MW, Goodnight WH, Tita ATN, Costantine MM, Swamy GK, Heyborne KD, Chien EK, Chauhan SP, El-Sayed YY, Casey BM, Parry S, Simhan HN, Napolitano PG, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units (MFMU) Network. Amniocentesis to diagnose congenital cytomegalovirus infection following maternal primary infection. Am J Obstet Gynecol MFM. 2022 Jul;4(4):100641. doi: 10.1016/j.ajogmf.2022.100641. Epub 2022 May 6. PMID 35526782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 206,082 Pregnant women were assessed for eligibility (screened for primary CMV infection). 205,683 Were excluded.
Period: Overall Study
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Started | 206 | 193
Completed | 203 | 191
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo | Total
Number analyzed (Participants) | 206 | 193 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (6.3) | 28.5 (6.0) | 27.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 193 | 399
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 135 | 124 | 259
  Non-Hispanic Black | 35 | 30 | 65
  Hispanic | 30 | 33 | 63
  Other, unknown, or more than one race or ethnic group | 6 | 6 | 12
Married or living with partner [Count of Participants; unit: Participants] | 145 | 142 | 287
Education [Mean (Standard Deviation); unit: years] | 14.1 (2.1) | 14.2 (2.3) | 14.2 (2.2)
Occupational exposure [Count of Participants; unit: Participants] — Includes teacher, student, babysitter or nanny, health care worker, or day-care worker. Population: Includes only participants who completed the self-report.
  Participants
    number analyzed (Participants) | 195 | 174 | 369
    (all) | 78 | 63 | 141
1 or more children living at home [Count of Participants; unit: Participants] | 150 | 140 | 290
1 or more children in day care [Count of Participants; unit: Participants] | 83 | 78 | 161
Nulliparous [Count of Participants; unit: Participants] | 75 | 62 | 137
Tobacco use [Count of Participants; unit: Participants] — Self-reported use of tobacco products
  Participants | 22 | 23 | 45
Alcohol use [Count of Participants; unit: Participants] — self-reported use of alcohol
  Participants | 21 | 24 | 45
CMV infection at screening [Count of Participants; unit: Participants] — One participant in the hyperimmune globulin group did not have primary cytomegalovirus (CMV) infection and underwent randomization in error.
  Participants
    IgM+, IgG+, low avidity (low avidity defined as less than 50 percent) | 200 | 183 | 383
    IgM+, IgG seroconversion | 5 | 10 | 15
    No primary CMV infection - randomization error | 1 | 0 | 1
Mean weeks gestation at randomization [Mean (Standard Deviation); unit: weeks] | 16.2 (3.9) | 15.6 (4.1) | 15.9 (4.0)
Distribution of weeks gestation at randomization [Count of Participants; unit: Participants]
  ≤11 weeks, 6 days | 26 | 36 | 62
  12 weeks, 0 days to 19 weeks, 6 days | 142 | 126 | 268
  ≥20 weeks, 0 days | 38 | 31 | 69
Body-mass index at randomization [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (7.0) | 26.9 (7.0) | 27.1 (7.0)
Avidity index at randomization [Mean (Standard Deviation); unit: avidity index] — Avidity is defined as the aggregate strength with which antibodies bind to antigen. Low avidity index is a reliable indicator of CMV infection within the previous 6 months, a high avidity index essentially excludes the possibility that infection occurred within the previous 4 months.
  Avidity index values are calculated on a 0% to 100% scale. Values less than 60% are interpreted as low avidity, and values greater than 70% are interpreted as high avidity; values from 60% to 70% (inclusive) are interpreted as intermediate avidity. Population: Data are not included for 4 participants (1 in the hyperimmune globulin group and 3 in the placebo group) who underwent seroconversion.
  avidity index
    number analyzed (Participants) | 205 | 190 | 395
    (all) | 29.7 (14.6) | 29.9 (13.6) | 29.8 (14.1)
Days from screening to randomization [Mean (Standard Deviation); unit: days] | 25.5 (9.1) | 25.2 (8.2) | 25.3 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Composite Primary Outcome
Description: The primary outcome is a binary outcome defined by the occurrence or non-occurrence of any of the following vs. none of the following: fetal loss (spontaneous or termination), confirmed fetal CMV infection from amniocentesis, neonatal death before assessment of CMV infection can be made, or neonatal congenital CMV infection. Neonatal congenital CMV infection is diagnosed by urine or saliva collected by 3 weeks of age that is positive for CMV by culture (the intent will be to obtain in the first two days of life). In the event that Polymerase Chain Reaction (PCR) is positive but culture is negative, a repeat culture must be positive by 3 weeks of age.
Time Frame: From randomization through 3 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 46 | 37
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; p = 0.42, Chi-squared; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.80 to 1.72]

2. Primary Outcome: Number of Participants Who Had a Fetus or Neonate With CMV Infection
Description: Component of composite primary outcome
Time Frame: From randomization through 3 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 36 | 32

3. Primary Outcome: Number of Participants Who Had a Neonatal Death Without CMV Infection
Description: component of composite primary outcome
Time Frame: From randomization through 3 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 0 | 0

4. Primary Outcome: Number of Participants With a Fetal or Neonatal Death With Proven CMV Infection
Description: component of primary composite outcome
Time Frame: From randomization through 3 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 7 | 3

5. Primary Outcome: Number of Participants With Fetal Death Without Proven CMV Infection
Description: component of primary composite outcome
Time Frame: From randomization through delivery
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 3 | 2

6. Secondary Outcome: Number of Participants With Gestational Hypertension or Preeclampsia
Description: Gestational hypertension or preeclampsia is a binary outcome defined by occurrence or non-occurrence of gestational hypertension or preeclampsia. Gestational hypertension or preeclampsia are new onset hypertension during pregnancy
Time Frame: from randomization through discharge from the hospital
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 205 | 193
Participants | 24 | 14
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.61, 95% CI 2-sided [0.86 to 3.03]

7. Secondary Outcome: Number of Participants With Placental Abruption
Description: Placental abruption is a binary outcome defined by occurrence or non-occurrence of placental abruption, defined as bleeding and contraction pain
Time Frame: From randomization through delivery (maximum 42 weeks gestation)
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 205 | 193
Participants | 3 | 1
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 2.82, 95% CI 2-sided [0.29 to 72.42]

8. Secondary Outcome: Median Gestational Age at Delivery
Description: Gestational age at delivery in weeks
Time Frame: Delivery
Measure: Median (Standard Deviation); unit: weeks
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
weeks | 38.2 (4.1) | 38.6 (3.6)
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Difference (RD) = -0.41

9. Secondary Outcome: Number of Participants Whose Gestational Age at Delivery Was Before 37 Weeks
Description: Gestational age before 37 weeks gestation is a binary outcome meaning occurrence or non-occurrence of delivery before 37 weeks gestation
Time Frame: Delivery before 37 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 25 | 16
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.47, 95% CI 2-sided [0.81 to 2.67]

10. Secondary Outcome: Number of Participants Whose Gestational Age at Delivery Was Before 34 Weeks, 0 Days
Description: Gestational age before 34 weeks, 0 days gestation is a binary outcome meaning occurrence or non-occurrence of delivery before 34 weeks gestation
Time Frame: Delivery before 34 weeks gestation
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 12 | 7
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.61, 95% CI 2-sided [0.65 to 4.01]

11. Secondary Outcome: Number of Participants Reporting Yes or no to Medication Side Effects
Description: Occurrence or non-occurrence of a designated side effect of medication
Time Frame: From randomization (10-27 weeks gestation) through delivery (maximum 42 weeks gestation)
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 206 | 193
Participants
  Participants reported no side effects | 125 | 131
  Participants reported any side effects | 81 | 62

12. Secondary Outcome: Number of Participants Who Had a Fetal or Neonatal Death
Description: Fetal death or death of a neonate born alive
Time Frame: From randomization (10-27 weeks gestation) through delivery (maximum 42 weeks gestation) up to 120 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 10 | 5
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.88, 95% CI 2-sided [0.66 to 5.41]

13. Secondary Outcome: Median Neonatal Head Circumference
Description: Neonatal head circumference measured within 72 hours of birth
Time Frame: 72 hours postpartum
Measure: Median (Standard Deviation); unit: centimeters
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
centimeters | 33.9 (2.1) | 34.1 (1.9)
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.66 to 0.15]

14. Secondary Outcome: Median Birth Weight
Description: Birth weight as recorded in the medical record
Time Frame: Delivery
Measure: Median (Standard Deviation); unit: grams
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
grams | 3268 (657) | 3303 (548)
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Difference (RD) = -35, 95% CI 2-sided [-157 to 87]

15. Secondary Outcome: Number of Participants With Fetal Growth Restriction
Description: Fetal growth restriction is a binary outcome defined as the occurrence or non-occurrence of growth restriction (defined as <5th percentile weight for gestational age, assessed specifically by sex and race of the infant based on United States birth certificate data)
Time Frame: Delivery
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 194 | 186
Participants | 20 | 10
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.92, 95% CI 2-sided [0.92 to 3.99]

16. Secondary Outcome: Number of Participants With Symptomatic CMV Infection
Description: Fetal or neonatal symptomatic CMV infection is a binary outcome defined as the occurrence or non-occurrence of symptomatic CMV infection defined as CMV isolated from an amniocentesis, or urine or saliva during the first three weeks of life and at least one of the following: jaundice (with direct bilirubin exceeding 20% of total bilirubin), thrombocytopenia , anemia , hepatitis, hepatomegaly, splenomegaly, growth restriction, failure to thrive, intracerebral calcifications, microcephaly, hypotonia, seizures, petechial rash, hearing loss, interstitial pneumonitis, thrombocytopenia, anemia, hepatitis, chorioretinitis, or CMV in cerebrospinal fluid
Time Frame: During pregnancy up to 3 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 203 | 191
Participants | 23 | 15

17. Secondary Outcome: Number of Neonates With Grade 3 or 4 Intraventricular Hemorrhage
Description: Intraventricular hemorrhage (IVH) as determined by cranial ultrasounds performed as part of routine clinical care and classified based on the Papile classification system. IVH is a binary outcome defined by occurrence or non-occurrence of IVH
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 1 | 0

18. Secondary Outcome: Number of Neonates With Ventriculomegaly
Description: Ventriculomegaly is a binary outcome defined by the occurrence or non-occurrence of ventriculomegaly
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 194 | 186
Participants | 1 | 0

19. Secondary Outcome: Number of Neonates With Retinopathy of Prematurity (ROP)
Description: Retinopathy of prematurity is a binary outcome defined by the occurrence or non-occurrence of retinopathy of prematurity, diagnosed by ophthalmologic examination of the retina and a diagnosis of Stage I (demarcation line in the retina) or greater.
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 1 | 1
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.03 to 31.5]

20. Secondary Outcome: Number of Neonates With Respiratory Distress Syndrome
Description: Respiratory distress syndrome is a binary outcome defined by the occurrence or non-occurrence of Respiratory distress syndrome (defined as the presence of clinical signs of respiratory distress (tachypnea, retractions, flaring, grunting, or cyanosis), with an oxygen requirement and a chest x-ray that shows hypoventilation and reticulogranular infiltrates).
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 5 | 10
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.48, 95% CI 2-sided [0.17 to 1.38]

21. Secondary Outcome: Number of Neonates With Chronic Lung Disease
Description: Neonatal chronic lung disease is a binary outcome defined by the occurrence or non-occurrence of chronic lung disease or bronchopulmonary dysplasia (BPD) defined as oxygen requirement at 28 days of life
Time Frame: 28 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 0 | 0

22. Secondary Outcome: Number of Neonates With Necrotizing Enterocolitis (NEC)
Description: Necrotizing enterocolitis (NEC) is a binary outcome defined by the occurrence or non-occurrence of NEC, defined as modified Bell Stage 2 or 3. Stage 2: Clinical signs and symptoms with pneumatosis intestinalis on radiographs. Stage 3: Advanced clinical signs and symptoms, pneumatosis, impending or proven intestinal perforation.
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 0 | 0

23. Secondary Outcome: Number of Neonates With Hyperbilirubinemia
Description: Hyperbilirubinemia is a binary outcome defined by the occurrence or non-occurrence of hyperbilirubinemia. Peak total bilirubin of at least 15 mg% or the use of phototherapy
Time Frame: From birth to 1 week of life
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 150 | 138
Participants | 13 | 19
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.63, 95% CI 2-sided [0.32 to 1.23]

24. Secondary Outcome: Number of Neonates With Suspected Neonatal Sepsis
Description: Suspected neonatal sepsis is a binary outcome defined as the occurrence or non-occurrence of suspected neonatal sepsis
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 14 | 16
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.42 to 1.68]

25. Secondary Outcome: Number of Neonates With Neonatal Pneumonia
Description: Neonatal pneumonia is a binary outcome defined as the occurrence or non-occurrence of neonatal pneumonia
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 1 | 2
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.47, 95% CI 2-sided [0.17 to 5.23]

26. Secondary Outcome: Number of Neonates Experiencing Seizures / Encephalopathy
Description: Neonatal seizures/encephalopathy is a binary outcome defined as the occurrence or non-occurrence of seizures/encephalopathy
Time Frame: 0 days to approximately 120 days of life or hospital discharge, whichever is sooner
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
Participants | 0 | 0

27. Secondary Outcome: Median Length of Neonatal Hospital Stay
Description: Length of hospital stay, need for Neonatal Intensive Care Unit (NICU) or intermediate care admission and length of stay if admitted
Time Frame: birth to neonatal hospital discharge (usually a maximum of 120 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 193 | 186
days | 2 [2 to 2] | 2 [2 to 2]

28. Secondary Outcome: Number of Participants Experiencing Infant or Child Death
Description: Death of infant or child before the 24 month study exam
Time Frame: Birth to 24 month study exam
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 184 | 176
Participants | 10 | 5

29. Secondary Outcome: Number of Children With Sensorineural Hearing Loss
Description: Sensorineural hearing loss is defined as the occurrence or non-occurrence of sensorineural hearing loss defined as unilateral and bilateral sensorineural hearing loss
Time Frame: 12 and 24 months corrected age
Population: Hearing data was not available for approximately 25% of children due to loss to followup or consent refusal.
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 138 | 146
Participants | 2 | 7

30. Secondary Outcome: Number of Children Diagnosed With Chorioretinitis
Description: Chorioretinitis is defined as the occurrence or non-occurrence of chorioretinitis defined by ophthalmologic exam
Time Frame: 2 years of age
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 173 | 171
Participants | 0 | 1

31. Secondary Outcome: Mean Cognitive Composite Scores From the Bayley Scales of Infant and Toddler Development Third Edition (Bayley-III)
Description: The Bayley Scales of Infant and Toddler Development® | Third Edition (Bayley®-III), is a comprehensive tool to identify development issues during early childhood. The Bayley-III Cognitive Scale subtests assess cognitive function through the use of memory, problem solving and manipulation subtests. Scores on individual Cognitive subtests range from 1 (worst outcome) to 19 (better outcome) (Mean 10, SD 3). Individual subtest scores between 8 and 12 are considered average. The raw scores on the subtests are converted to scaled scores based on American norms by age. Cognitive Scale composite scores range from 55 (low, worse outcome) to 155 (high, better outcome) (mean 100; SD 15). Severe disability was defined as a composite score <70.
Time Frame: 12 and 24 months corrected age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 155 | 160
score on a scale | 96.2 (15.1) | 97.1 (13.5)

32. Secondary Outcome: Mean Motor Composite Scores From the Bayley Scales of Infant and Toddler Development Third Edition (Bayley-III)
Description: The Bayley Scales of Infant and Toddler Development® | Third Edition (Bayley®-III), is a comprehensive tool to identify development issues during early childhood. The Bayley-III Motor Scale subtests assess motor function through fine motor and gross motor subtests. Scores on individual Motor subtests range from 1 (worst outcome) to 19 (better outcome) (Mean 10, SD 3). Individual subtest scores between 8 and 12 are considered average. The raw scores on the subtests are converted to scaled scores based on American norms by age. Motor Scale composite scores range from 55 (low, worse outcome) to 155 (high, better outcome) (mean 100; SD 15). Severe disability was defined as a composite score <70.
Time Frame: 12 and 24 months corrected age
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 155 | 158
score on a scale | 98.7 (16.4) | 101.9 (14.9)

33. Secondary Outcome: Number of Infants or Children With the Composite Outcome
Description: Composite outcome at 24 months including any of the following attributable to congenital CMV infection: • Sensorineural hearing loss (unilateral and bilateral) • Developmental delay defined as Cognitive score < 70 or Motor score < 70 on the Bayley III • Chorioretinitis • Fetal loss or death of neonate, infant or child
Time Frame: 24 month study exam
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 149 | 149
Participants | 20 | 15
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; p = 0.37, Chi-squared; Risk Ratio (RR) = 1.3, 95% CI 2-sided [0.7 to 2.5]

34. Secondary Outcome: Overall Child Status at 24 Months of Age
Description: Child status at age 24 months, classified as: • Fetal loss or death of neonate, infant or child • Congenital CMV infection with severe disability • Congenital CMV infection without severe disability • Infant not infected with CMV
Time Frame: 24 month study exam
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 148 | 149
Participants
  Death or fetal loss | 10 | 5
  Congenital CMV with severe disability | 6 | 7
  Congenital CMV without severe disability | 21 | 19
  Not infected with CMV with severe disability | 4 | 3
  Not infected with CMV and no disabilities | 107 | 115
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; p = 0.26, Chi-squared

35. Secondary Outcome: Failure to Thrive at 24 Months
Description: Failure to thrive defined as <10th percentile for weight at 24 months
Time Frame: 24 months of age
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
Number analyzed (Participants) | 169 | 167
Participants | 20 | 21
Statistical Analysis 1: Comparison: CMV Hyperimmune Globulin - Cytogam® vs Placebo; Test type: Superiority; p = 0.84, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected from randomization through delivery (a time period of up to 36 weeks)
Description: Adverse events are described in general terms and grouped where possible to protect the confidentiality of participants, given that some events rarely occurred.
Arm/Group | CMV Hyperimmune Globulin - Cytogam® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/193
Serious Adverse Events (participants affected / at risk) | 32/206 | 25/193
Other Adverse Events (participants affected / at risk) | 8/206 | 7/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMV Hyperimmune Globulin - Cytogam® (N=206) | Placebo (N=193)
hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Congenital Anomaly (Congenital, familial and genetic disorders) | 9 (9) | 2 (2)
Serious allergic reaction (General disorders) | 2 (2) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Corpus callosum lesion (Nervous system disorders) | 0 (0) | 1 (1)
Elective termination (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 2 (2)
Fetal death (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3)
Preterm birth (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 10 (10)
Respiratory syncytial virus (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Meconium aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMV Hyperimmune Globulin - Cytogam® (N=206) | Placebo (N=193)
congenital anomaly (non-serious) (Congenital, familial and genetic disorders) | 5 (5) | 5 (5)
allergic reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT01376778/Prot_SAP_ICF_000.pdf